CLINICAL TRIAL: NCT03534089
Title: Effectiveness of the Treatment for Infant Iron Deficiency Anemia by Taking Lactoferrin and Ferralia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beingmate Baby & Child Food Co Ltd . (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RD07316001A
Record Dates: First submitted 2018-04-27; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2017-12

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard infant fomula (Placebo Comparator): Infants with iron deficiency anemia randomly divided into this arm were given the same dose of ferralia with other arms,but were fed with standard infant formula (without lactoferrin supplementation)
  Interventions: Other: Standard infant fomula
- Low level LF infant formula group (Experimental): Infants with iron deficiency anemia randomly divided into this arm were given the same dose of ferralia with other arms,but were fed with infant formula supplemented with low level of lactoferrin (38mg/100g). Lactoferrin:38mg/100g
  Interventions: Other: Low level LF infant formula
- High level LF infant formula group (Experimental): Infants with iron deficiency anemia randomly divided into this arm were given the same dose of ferralia with other arms,but were fed with infant formula supplemented with high level of lactoferrin (76mg/100g)
  Interventions: Other: High level LF infant formula

INTERVENTIONS:
Other: Standard infant fomula — Infants with iron deficiency anemia randomly divided into this group were given the same dose of ferralia with other groups,and were fed with infant formula without lactoferrin supplementation.
  Arms: Standard infant fomula
Other: Low level LF infant formula — Infants with iron deficiency anemia randomly divided into this group were given the same dose of ferralia with other groups,and were fed with infant formula supplemented with low level of lactoferrin (38mg/100g).
  Arms: Low level LF infant formula group
Other: High level LF infant formula — Infants with iron deficiency anemia randomly divided into this group were given the same dose of ferralia with other groups,and were fed with infant formula middle supplemented with high level of lactoferrin (76mg/100g).
  Arms: High level LF infant formula group

SUMMARY:
A multi-center,randomized,double-blind,controlled clinical trial was used to investigate the effectiveness of the treatment of infant iron deficiency anemia by taking ferralia and different contents lactoferrin.

DETAILED DESCRIPTION:
5-9 months old infants with iron deficiency anemia were randomly divided into three groups. On the basis of giving the same dose of ferralia,three different levels lactoferrin infant formula were intervened 3 months respectively,and evaluate the clinical effect.

ELIGIBILITY:
Inclusion Criteria:

* Full term,healthy infants at 37-42 weeks of gestational age
* 5-9 months old infants were diagnose as iron deficiency anemia
* Accepting bottle feeding

Exclusion Criteria:

* Hb<60 g/L
* Other microcytic, hypochromic anemia

Ages: 5 Months to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Changes of Hb concentration(g/L) | Change of Hb concentration from baseline at 1 month and 3 months.
  Hb was measured by the hemoglobincyanide method

SECONDARY OUTCOMES:
Change of body weight (kilograms) | Changes of body weight from baseline at 1 month and 3 months.
  Body weight is detected by electronic scale
Change of body length (meters) | Changes of body weight from baseline at 1 month and 3 months.
  Body length is detected by infant height bed
Change of head circumference (millimeters) | Changes of body weight from baseline at 1 month and 3 months.
  Head circumference detected by measuring tape
Change of serum ferritin concentration (μg/L) | Changes of serum iron concentration from baseline at 3 months.
  concentrations of serum ferritin (SF,μg/L) were measured using a commercial enzyme-linked immunosorbent assay (ELISA; Sunbiote, Shanghai, China).
Change of serum transferrin receptor concentration(mg/L) | Changes of serum transferrin receptor concentration from baseline at 3 months.
  Serum soluble transferrin receptor (sTfR, mg/L) was measured by microparticle-enhanced immunoassay (Sunbiote, Shanghai, China)

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Women's and Children's Central Hospital, Chengdu, China